CLINICAL TRIAL: NCT01388322
Title: Enoxaparin for the Prevention of Placental-Mediated Complications of Pregnancy in Women With Obstetric History or Abnormal Uterine Artery Doppler at First Trimester Ultrasound and Without Thrombophilia: a Multicenter Randomized Controlled Trial
Brief Title: Low Weight Heparin prOphylaxis for Placental-Mediated Complications of PrEgnancy
Acronym: HOPPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Hospital Vall d'Hebron (Other); Hospital Sant Joan de Deu (Other); Hospital de Cruces (Other); Parc Sanitari Sant Joan de Déu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HOPPE-Trial; 2010-023597-39 (EudraCT Number)
Record Dates: First submitted 2011-06-28; First posted 2011-07-06 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: High Risk Pregnant Women; Placental Insufficiency; Preeclampsia
Keywords: Pregnancy; Preeclampsia; Placental insufficiency
MeSH Terms: conditions — Placental Insufficiency; Pre-Eclampsia | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enoxaparin (Experimental): Subcutaneous administration of one dose daily of enoxaparin
  Interventions: Drug: Enoxaparin
- expectant management (No Intervention): Usual management

INTERVENTIONS:
Drug: Enoxaparin — 40 mg (4000 IU) women <80 kg at the time of randomization or 60 mg (6000 IU) women> 80 kg at the time of randomization One dose daily. Subcutaneous administration. Treatment periods: the same day of the Initiation visit (from 9 to 13.6 weeks of gestation) until 36 weeks gestation.
  Arms: Enoxaparin

SUMMARY:
This is a Multicenter, randomized, open-label, parallel groups study to test the hypothesis that prophylactic low molecular weight heparin (LMWH) (enoxaparin) initiated before 14 weeks of gestation could improve maternal and perinatal outcome in women at high risk for developing placental-mediated pregnancy complications.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ≥18 years
* Gestational age < 14 weeks at randomisation
* One or more of the following complications in a previous pregnancy:

  * Severe PE resulting in delivery before 32 weeks of gestation
  * Newborn weight less than the 10th percentile and documented abnormal Doppler in the umbilical artery during pregnancy before 32 weeks gestation
  * Abruption of placenta
  * Unexplained intrauterine death between 20-41,6 weeks of gestation secondary of placental insufficiency or
* Uterine arteries Pulsatility Index (mPI) Doppler ≥95th percentile at 11-14 weeks of gestation.

Exclusion Criteria:

* Multiple pregnancy
* Abnormal thrombophilia study
* Alcohol or illicit drug use
* Severe fetal malformations or chromosomal abnormalities
* Previous history of infertility ( 3 or more early miscarriages)
* Maternal HIV, Cytomegalovirus or toxoplasma infection
* Known fetal abnormality or chromosomal defect at randomisation
* Women with previous venous or arterial thrombotic event
* Organic lesions that could increase the hemorrhagic risk: gastric ulcus, stroke, a recent hemorrhagic event, high risk situations for hemorrhagic event
* Known allergy to heparin or LMWH, thrombopenia or thrombosis episode due to heparin treatment
* Contraindication to LMWH
* An absolute indication for anticoagulant therapy: venous deep thrombosis, pulmonary embolism, ovaric hyperestimulation, cardiophaty, others
* Metabolic disorders a risk for development of PE and/or IUGR: Type I diabetes, hipertiroidism, chronic renal insufficiency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Estimated)
Dates: Start 2012-03; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Development of any of these complications of placental insufficiency | from date of randomization until the date of delivery (assessed up to 30 weeks)
  Development of any of these complications of placental insufficiency: preeclampsia, intrauterine growth restriction, abruption placentae, and/or intrauterine fetal demise

SECONDARY OUTCOMES:
Gestational age at birth | from date of randomization until the date of delivery (assessed up to 30 weeks)
  Gestational age at birth
Days of hospitalization during pregnancy | from randomization to the time of delivery (30 weeks)
  Days of hospitalization during pregnancy
Days of maternal hospitalization in the postpartum period | from delivery until discharge (an expected average of one week)
  Days of maternal hospitalization in the postpartum period
Neonatal Data | after the delivery (an expected average of one month)
  weight, height, head circumference, Apgar score 1-5 min, arterial pH, venous base excess (BE) of umbilical cord gases, and complications

CONTACTS AND LOCATIONS:
Overall Officials: Lluís Cabero, MD PhD, Study Chair — Hospital Vall d'Hebron; Elisa Llurba, MD, Principal Investigator — Hospital Vall d'Hebron; Maria Dolores Gómez, MD, Principal Investigator — Hospital Sant Joan de Deu; Txantón Martínez-Astorquiza, MD, Principal Investigator — Hospital de Cruces; Raul De Diego, M.D., Principal Investigator — Parc Sanitari Sant Joan de Deu
Locations (4):
- Spain (4):
  - Hospital Universitario Vall d'Hebron, Barcelona, Barcelona
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Parc sanitari Sant Joan de Deu, Sant Boi de Llobregat, Barcelona
  - Hospital de Cruces, Barakaldo, Vizcaya